CLINICAL TRIAL: NCT05450497
Title: Effect of Propofol vs Dexmedetomidine or Propofol+Dexmedetomidine on Reducing the Frequency of Arrhythmia in Patients After Cardiac Surgery
Brief Title: Effect of Sedative Agent on Reducing the Frequency of Arrhythmia in the Patients After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anesthesia Research Group UA (Other)
Responsible Party: Principal Investigator, Plechysta Yelyzaveta, Chief of the anesthesia Department, Anesthesia Research Group UA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0120U100655
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Arrythmia
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Propofol Group (Experimental): Patient sedation after cardiac surgery at the intensive care unit. Continuous infusion of propofol using a syringe pump at the dose of 1-1.5 mg / kg / h
  Interventions: Drug: Propofol
- Dexmedetomidine (Experimental): Patient sedation after cardiac surgery at the intensive care unit. Continuous infusion of Dexmedetomidine using a syringe pump at the dose of 0.5-1.0 mcg/ kg / h
  Interventions: Drug: Dexmedetomidine
- Dexmedetomidine and propofol (Experimental): Patient sedation after cardiac surgery at the intensive care unit.
  Sedation group DEX+PR:
  continuous infusion of propofol using a syringe pump at the dose of 0.5-1.5 mg / kg / h and dexmedetomidine 0.2-0.7 mcg\kg\h
  Interventions: Drug: Dexmedetomidine and propofol

INTERVENTIONS:
Drug: Propofol — comparing sedative agents
  Arms: Propofol Group
Drug: Dexmedetomidine — comparing sedative agents
  Arms: Dexmedetomidine
Drug: Dexmedetomidine and propofol — comparing sedative agents
  Arms: Dexmedetomidine and propofol

SUMMARY:
Arrhythmias early in the recovery period after cardio thoracic surgery are common they develop in 11 to 40 percent of patients after coronary-artery bypass grafting. The right chose of sedative agent could decrease the level of arrhythmia incidence.

DETAILED DESCRIPTION:
Arrhythmias are really common in patients after cardiac surgery. Most of the patients get sedation after cardiac surgery. The goal is to determine if the propofol (PR) (sedative agent), dexmedetomidine (DEX)(selective α2-adrenergic receptor (α2-AR) agonist) or their combination could improve and decrease the incidence of the arrhythmia in patients after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Multi vascular lesions of the coronary arteries according to coronary angiography;
* Heart valve damage was confirmed by heart ultrasound, which is subject to surgical correction (aortic stenosis of III degree with a gradient on the aortic valve of more than 42 mmHg, aortic insufficiency III, mitral valve stenosis II-III, mitral regurgitation II-III)
* Age of patients from 18-80 years;

Exclusion Criteria:

* Refusal to participate;
* Hypersensitivity to propofol, dexmedetomidine;
* Acute renal failure that occurred during surgery (ClCr less than 50 ml / h, or a decrease in the rate of diuresis to 0.1 ml / h in the first 4 hours after surgery and does not respond to diuretic therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
incidence of arrhythmia | day of the discharge from the hospital (assessed up to day 5)
  incidence of deviation from the rhythm before the surgery and at the day of the discharge from the hospital after cardia surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yelyzaveta Plechysta, MD, Study Chair — Chief of the anesthesia department
Locations (1):
- Medical Network Dobrobut, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No